CLINICAL TRIAL: NCT03998228
Title: Association Between Dermatoporosis and Fractural Risk
Acronym: DermatOstéo
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: TSE_2019_11
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-11

CONDITIONS: Dermatoporosis
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual X-ray absorptiometry (DMO) densitometry. — Simple clinical examination with forearm inspection and palpation;
  * Radiological examination of BMD;
  * Calculation of the FRAX® score;
  * Fact sheet on patients with dermatoporosis, proposal of a topical treatment (cosmetic cream) and completion of the questionnaire specific to dermatoporosis

SUMMARY:
There is a need for new tools to identify patients who may have osteoporosis before a fracture occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 40 and 90 years old who has to undergo a bone densitometry (BMD) examination by dual X-ray absorptiometry
* Affiliate or beneficiary of a Social Security scheme
* Express consent to participate in the study.

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or nursing woman.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients who are to perform dual X-ray absorptiometry (DMO) densitometry.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
compare fracture risk between patients with dermatoporosis and those without dermatoporosis | BASELINE
  The fracture risk will be calculated using the FRAX score. The presence of dermatoporosis will be assessed by a simple clinical examination of the forearms and defined by the presence of three clinical signs: cutaneous atrophy, Bateman purpura and presence of pseudo-stellar scars.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SENE, MD PhD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No